CLINICAL TRIAL: NCT00925730
Title: Non-comparative Open-label Study to Investigate the Efficacy, Safety and Systemic Exposure of Pimecrolimus in Adult and Pediatric Patients With Moderate to Severe Atopic Dermatitis Treated Topically for 8.5 Days With Pimecrolimus Cream 1% Under Occlusion
Brief Title: Open-label Study to Investigate Systemic Exposure in Adult and Pediatric Atopic Dermatitis Patients Treated 8.5 Days With Pimecrolimus Cream 1% Under Occlusion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASM981C2313
Record Dates: First submitted 2009-06-17; First posted 2009-06-22 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Atopic Dermatitis
Keywords: Atopic dermatitis; AD; pimecrolimus; blood; absorption; systemic
MeSH Terms: conditions — Dermatitis, Atopic | interventions — pimecrolimus

ARMS (1):
- Pimecrolimus cream 1% (Experimental): Pimecrolimus
  Interventions: Drug: Pimecrolimus

INTERVENTIONS:
Drug: Pimecrolimus

SUMMARY:
This study will access the degree to which pimecrolimus is absorbed from pimecrolimus cream 1% into the blood when applied repeatedly under occlusion (i.e. areas treated wrapped in a plastic film) over 8 days in patients with moderate to severe atopic eczema.

ELIGIBILITY:
Inclusion Criteria:

* Patients 2 - 18 years of age
* Patients with a diagnosis of moderate to severe atopic dermatitis, assessed by a score ≥ 3 at the Investigator's Global Assessment. AD to involve at least 30% of their body surface area as determined by the rule of nine or the Lund and Browder chart.

Exclusion Criteria:

* Erythrodermic patients with Netherton's syndrome
* Patients with known serious adverse reactions or hypersensitivity to any of the excipients of the study medication
* Patients with a history of cancer, skin malignancy or lymphoproliferative disorders or of immunocompromise, including a positive HIV (ELISA and Western blot), Hepatitis B surface antigen (HBsAg) or Hepatitis C test result

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2004-03; Primary Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Pimecrolimus blood concentration | Days 1, 9, 16

SECONDARY OUTCOMES:
Efficacy as assessed by the Eczema Area and Severity Index and the Investigators Global Assessment of disease severity. Efficacy outcomes were of an exploratory nature in this study. | Days 1, 9, 16

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Germany (2):
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Frankfurt am Main

REFERENCES:
- [Result] Thaci D, Kaufmann R, Bieber T, Hanfland J, Hauffe S, Koehne-Voss S, Waldmeier F. Percutaneous absorption of pimecrolimus is not increased in patients with moderate to severe atopic dermatitis when pimecrolimus cream 1% is applied under occlusion. Dermatology. 2010;221(4):342-51. doi: 10.1159/000320125. Epub 2010 Nov 22. PMID 21099191